CLINICAL TRIAL: NCT00826891
Title: Phase II Study of Cisplatin Combined With Topotecan in Advanced (Stage IVB) Recurrent or Persistent Cervical Cancer
Brief Title: Study of Cisplatin in Cervical Cancer Stage IVB
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Anti-Cancer Association (Other)
Responsible Party: xuan guo, Chinese Anti-Cancer Association
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CACA-2008-GSK1
Record Dates: First submitted 2009-01-16; First posted 2009-01-22 (Estimated); Last update posted 2009-01-22 (Estimated); Status verified 2009-01

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Topotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cisplatin Combined With Topotecan — Patients must have specific minimum neutrophil and platelet counts before administration of Hycamtin. The dose of Hycamtin is 0.75 mg/m2 by intravenous infusion over 30 minutes daily on days 1, 2, and 3; followed by cisplatin 50 mg/m2 by intravenous infusion on day 1 repeated every 21 days (a 21-day course).
  Dosage adjustments for subsequent courses of Hycamtin in combination with cisplatin are specific for each drug.
  Dose levels for cisplatin Initial dose 0 = 50 mg/m2 Dose reduction level -1 = 37.5 mg/m2 Dose reduction level -2 = 25 mg/m2
  Dose levels for topotecan Initial dose 0 = 0.75 mg/m2 Dose reduction level -1 = 0.60 mg/m2 Dose reduction level -2 = 0.45 mg/m2

SUMMARY:
This is a single arm, open-label study in women from China who have Advanced (stage IVB) Recurrent or Persistent cervical cancer to ⑴assess the response rate (i.e., CR + PR) of Cisplatin combined with Topotecan in treatment of advanced (stage IVB) recurrent or persistent Cervical cancer; ⑵assess the toxicities of CT regimen in treatment of cervical cancer. Prior to treatment, written informed consent should be obtained from all patients. Eligible patients will be assigned to CT regimen. The CT regimen is topotecan 0.75 mg/m2 IV during 30minutes days 1, 2, and 3; followed by cisplatin 50 mg/m2 IV on day1, repeated every 21 days. The study will consist of two phases: the safety run-in phase and study phase.

ELIGIBILITY:
Inclusion Criteria:

* women with advanced recurrent or persistent carcinoma of the uterine cervical who were unsuitable candidates for curative treatment with surgery and/or radiotherapy.
* Histologic types included squamous, adenosquamous, and adenocarcinoma of the cervia.
* Patients must be at least 18 years old.
* Measurable and/or evaluable disease parameters will be documented and recorded using clinical evaluation (and using CT for pathologic nodes when present).
* Life expectation greater than 3 months.
* Patients must have adequate organ function.
* Patients without history of sensitivity to camptothecin or platinum.
* Patients who are non-child-bearing potential, or consistent and correct use of methods of birth control from 2 weeks prior to administration of the first dose of study medication until 28 days after the final dose of observational medication.
* performance status 0 to 2; to have recovered from the effects of recent surgery, chemoradiotherapy, or radiotherapy; and to be free of clinically significant infection.
* Written informed consent

Exclusion Criteria:

* Patients with uncontrolled infections.
* Patients with concurrent severe medical problems unrelated to the malignancy which would expose the patient to extreme risk.
* Patients who received another investigational drug within 30 days prior to study entry.
* Patients who are receiving concurrent other chemotherapy, hormonal, immunotherapy or radiotherapy. Radiotherapy for palliation of related bone metastases is permitted.
* Patients with a history of allergic reactions to compounds chemically related to topotecan or platinum.
* Patients who are pregnant or lactating
* Concomitant malignancies or previous malignancies within the last five years, with the exception of adequately treated basal or squamous cell carcinoma of the skin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-01 (Estimated); Study Completion 2010-01 (Estimated)

PRIMARY OUTCOMES:
Response rate (CR + PR) (RECIST) | 4~6 weeks after the end of treatment

SECONDARY OUTCOMES:
Toxicity [NCI CTCAE (Version 3.0)] | 4~6 weeks after the end of treatment